CLINICAL TRIAL: NCT06833281
Title: An Open-label Extension of SPG302-ALZ-101 Study to Evaluate the Long-term Safety and Efficacy of Daily Oral SPG302 Treatment in Participants With Mild-to-Moderate Alzheimer's Disease (AD)
Brief Title: Extension Study of Participants From SPG302-ALZ-101
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: patients treated on compassionate use program
Sponsor: Spinogenix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPG302-ALZ-102 OLE
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; synapse; neural connectivity
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Open Label extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label Extension (Experimental): Active SPG302 to be administered to adult participants with AD who completed initial study. Dose to be administered to be dose received during previous study.
  Interventions: Drug: SPG302

INTERVENTIONS:
Drug: SPG302 — small synthetic molecule

SUMMARY:
This study will evaluate the long-term safety and efficacy of participants enrolled in SPG302-ALZ-101 with mild to moderate Alzheimer's Disease (AD)

DETAILED DESCRIPTION:
This is an open-label extension study of SPG302-ALZ-101 to investigate the long-term safety, tolerability, and efficacy of SPG302 administered orally in participants with mild-to-moderate AD. Enrolled participants will continue at the dose they received at the end of the first trial, and will self-administer SPG302 orally every day for up to 52 weeks. Participants will have an in-person clinic visit every 3 months (± 3 days) and a monthly phone visit. An end of treatment visit will occur within 7 days of the last dose of SPG302. A final visit to collect safety data will be conducted up to 1 month (± 3 days) post last dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate AD
* Clinical laboratory values within normal range or < 1.5 times ULN
* Life expectancy of >2 years
* Able and willing to provide written informed consent
* Must have participated in all study activities of SPG302-ALZ-101, the parent study

Exclusion Criteria:

Any physical or psychological condition that prohibits study completion

* Known cardiac disease
* Active or history of malignancy in the past 5 years
* Serious infection that will not be resolved by first day of study intervention.
* History of clinically significant CNS event or diagnosis in the past 5 years.
* Acute illness within 30 days of Day 1
* History of suicidal behavior or suicidal ideation
* History of chronic alcohol use or substance abuse in the last 5 years
* HIV, hepatitis B and/or hepatitis C positive
* Vaccines within 14 days
* Receipt of investigational products within 30 days
* Blood donation within 30 days
* Pregnant or breastfeeding

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events and serious adverse events | Up to 52 weeks
  Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)
C-SSRS (Columbia Suicide Severity Rating Scale) | Up to 52 weeks
  Prospective suicidality assessment is performed using the Columbia-Suicide Severity Rating Scale (C-SSRS), a questionnaire to evaluate suicidal ideation and behavior. Answer "yes" on item 4 or 5 of the Suicidal Ideation section or "yes" on any item of the Suicidal Behavior section is considered positive. The suicidal behavior lethality sub-scale evaluates the level of actual or potential medical damage. The range is 0-25.Min is 0 and Max is 25.

SECONDARY OUTCOMES:
Change in Mini-Mental State Examination (MMSE) from baseline to endpoint | up to 52 weeks
  The Mini-Mental State Exam (MMSE) is a test of cognitive function. It includes tests of orientation, attention, memory, language and visual-spatial skills. The lower the score the greater the impairment. The range is 0-30. Min is 0 and Max is 30.
Change in Alzheimer's Disease Assessment Scale-Cog (ADAS-COG) total score from baseline to endpoint | up to 52 weeks
  The ADAS-COG measures language and memory, focusing on cognitive and non-cognitive functioning. It evaluates word recall, naming of objects, word recognition, comprehension and word finding. The ADAS-COG is scored 0-70. Min is 0 and Max is 70. The higher the score the greater the impairment.
Quality of Life in Alzheimer's Disease (QOL-AD) from baseline to endpoint | up to 52 weeks
  The QOL-AD is a test to evaluate the quality of life through a series of questions of ability to complete daily activities and tasks. A lower score indicates lower functional quality of life. Per question scored at 1-2-3-4. Overall range is Min is 13 and Max is 52.
Change in Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS - CGIC) from baseline to endpoint | up to 52 weeks
  The ADCS - CGIC is a metric for clinical assessment of symptom severity. It consists of 2 parts. First a baseline evaluation of patient and caregiver is performed to collect necessary clinical information. The clinician will then conduct the second phase of the assessment after a specified time period, and changes in symptom severity are indicated on a seven-point scale. A higher scale indicates a worsening of symptoms. Range is 1-7. Min 1 and Max is 7.
Change in Alzheimer's Disease Clinical Dementia Rating Sum of Boxes (CDR-SB) from baseline to endpoint | up to 52 weeks
  The CDR-SB is an interview performed with patient and caregiver, and will stage the severity of cognitive impairment. The higher the score, the greater the impairment. Range is 0-18. Min is 0 and Max is 18.
Change in Alzheimer's Disease Cooperative Study - Daily Living Inventory (ADCS-ADL) from baseline to endpoint. | up to 52 weeks
  The ADCS-ADL is a metric to assess the ability to perform basic and instrumental activities of daily living. It is completed by a caregiver as a questionnaire or interview questions, and evaluates activities within the previous four weeks. Changes in symptom severity are indicated on a seven-point scale. A lower scale indicates greater impairment. Each question is 0-3. Total score is 78. Min is 0 and Max is 78.
Change in serum neurofilament light chain (NfL) in participants with AD from baseline to endpoint. | up to 52 weeks
  To assess the effect of SPG302 on Neurofilament light (NfL), a protein elevated in AD. This will be measured in picometers/milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Priest, MBBS, Principal Investigator — Flinders Medical Center, Adelaide, SA, Australia; Brew Brew, MBBS, MD, DSC, Principal Investigator — St Vincents Hospital, Sydney, NSW, Australia
Locations (2):
- Australia (2):
  - St. Vincent's Hospital, Sydney, New South Wales
  - Flinders Medical Center, Adelaide, South Australia